CLINICAL TRIAL: NCT01013441
Title: Trial of Immune Reconstitution With CD3/CD28 Bead Activated T-Cells Following Chemo-Immunotherapy in Patients With Chronic Lymphocytic Leukemia
Brief Title: CD3/CD28 Bead Activated T-Cells Following Chemo-Immunotherapy in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 15408; NCT00870090 (obsolete NCT alias)
Record Dates: First submitted 2009-11-05; First posted 2009-11-13 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Biological: Infusion of CD3/CD28 stimulated T cells

INTERVENTIONS:
Biological: Infusion of CD3/CD28 stimulated T cells — Receive CD3/CD28 stimulated T cells after fludarabine or alemtuzumab based chemotherapy
  Other Names: Activated T cells; CD3/CD28 stimulated T cells; T cells

SUMMARY:
The purpose of this research study is to test whether giving T-cells (type of white blood cell that are also known as immune cells) that have been specially processed in the laboratory will help chronic lymphocytic leukemia (CLL) patients' immune system return to normal faster after chemotherapy. This research study will also look into the ability of the lab to process the T-cells for infusion and the side effects of giving T-cells to patients with chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
Single arm, multi-center trial to evaluate the efficacy of administering CD3/CD28 stimulated T cells to chronic lymphocytic leukemia (CLL) patients following treatment with fludarabine or alemtuzumab based chemo- immunotherapy. All patients will undergo an apheresis to collect peripheral blood mononuclear cells (PBMCs) for generation of expanded T cells post- chemo-immunotherapy. Those subjects who achieve a complete or partial response to the chemoimmunotherapy based regimen will receive an infusion of 1.0 x 1010 (+/- 20%) activated autologous T cells expanded from the collected apheresis unit. Prior to T-cell infusion, at Day +30, +60, and +365 after T cell infusion, blood draws will be performed to assess immune reconstitution and immune function as compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL by immunophenotyping and flow cytometry analysis of blood or bone marrow.
* Patients with Rai stage III-IV - OR - Patients with Rai stage 0-II
* Zubrod performance status of 0-3
* Prior treatment with fludarabine or alemtuzumab based regimens.
* No untreated or uncontrolled life-threatening infection
* Women of childbearing potential must have a negative serum pregnancy test and agree to use a medically accepted form of contraception from the time of initial screening through completion of the study
* No active CNS disease
* Negative tests for HIV antibodies, Hepatitis B surface antigen, and hepatitis C antibodies.

Exclusion Criteria:

* Receipt of glucocorticoids (with the exception of inhaled glucocorticoid steroids for the use of allergic rhinitis or pulmonary disease) within 2 months prior to registration
* History of autoimmune disease unrelated to CLL (e.g., rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosis). Autoimmune disease related to CLL, e.g.

idiopathic thrombocytopenic purpura (ITP) or autoimmune hemolytic anemia, is permitted if not requiring active treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The occurrence of treatment-related adverse events or treatment related trial discontinuations, defined as NCI CTC ≥ grade 3 and clinical events that are possible, likely, or definitely related to study treatment at any time | Two years
The ability to complete the outlined course of therapy | Two years
The ability to harvest, expand, and reinfuse autologous T cells in this target population of patients | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Schuster, MD, Principal Investigator — Abramson Cancer Center, University of Pennsylvania; Chitra Hosing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Abramson Cancer Center, University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, University of Texas, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org/
- See also: Abramson Cancer Center — http://www.penncancer.org/